CLINICAL TRIAL: NCT02912897
Title: An Open Single-center, Phase I Proof of Concept Trial to Assess the Safety and Feasibility of Adoptive Cell Therapy with Autologous EBV-specific Cytotoxic T Lymphocytes (CTL) in Patients with a First Clinical Episode Highly Suggestive of Multiple Sclerosis
Brief Title: Trial to Assess the Safety and Feasibility of Adoptive Cell Therapy with Autologous EBV-specific Cytotoxic T Lymphocytes (CTL) in Patients with a First Clinical Episode Highly Suggestive of Multiple Sclerosis
Acronym: MS and EBV-CTL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC14_0359
Record Dates: First submitted 2016-09-13; First posted 2016-09-23 (Estimated); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis
Keywords: EBV-CTL; Multiple sclerosis; cellular therapy
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cellular therapy with EBV specific autologous CTL infusion (Experimental)
  Interventions: Biological: Cellular therapy with EBV specific autologous CTL infusion

INTERVENTIONS:
Biological: Cellular therapy with EBV specific autologous CTL infusion — CTL infusions at D0, M3 and M6

SUMMARY:
The etiologic mechanisms involved in multiple sclerosis (MS) are not yet fully understood. Indeed MS is a multifactorial disease involving genetic and environmental factors and Epstein-Barr-Virus (EBV) could be one of these factors. However the link between EBV infection and the immunological mechanisms underlying MS is not clear. Robust sero-epidemiological evidences support an association between EBV infection and MS, and immunological data suggest an altered/deficient immune response against this virus. In healthy individuals EBV produces a persistent infection that is tightly controlled by the immune system. In patients with MS, cellular and humoral immune studies demonstrate an altered response against the virus with a T-cell abnormal reactivity against the EBV-infected autologous B-cells, elevated humoral immune response to Epstein Barr Nuclear Antigen-1, and in the case of children, an increased EBV shedding, demonstrating frequent EBV reactivations. Thus, it has been proposed, that patients with MS present a partially inefficient control of the EBV infection. Some experimental data support the hypothesis suggesting that the presence of autoreactive EBV-B cells in the meninges of patients, probably due to an insufficient clearance of these cells by the immune system, lead to the infiltration of autoreactive T cells. Another hypothesis also suggests a deficient control of the virus, in that case during the inactive phase of the disease. Together, the above data and hypotheses lead to the notion that an immune intervention capable of restoring the host-EBV balance could be beneficial to MS patients In this project, we will assess the feasibility and safety of autologous transfer of several amounts of CD8 T cells directed against autologous EBV transformed B cell lines, in order to finally restore an efficient control of EBV in MS patients. The main objective of the project is to test the feasibility and safety of the process, while efficacy parameters will be also assessed in secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* 18<Age≤45 years
* Patients with :

  * A clinically isolated syndrome (first acute or sub acute neurological event consistent with demyelination [i.e. optic neuritis, spinal cord syndrome, brainstem/ cerebellar syndrome])
  * And a MRI scan showing dissemination of MRI lesions in space based on 2017 McDonald criteria At least 1 lesion detected in 2 or more following locations (sites) periventricular, cortical or juxtacortical, infratentorial, spinal cord
  * With a possible dissemination in time based on the revised McDonald cirteria and evicenced on simultaneous detection of one Gadolinium (Gd) enhancing and non-Gd enhancing lesions
  * Or demonstration of CSF-specific oligoclonal bands (OCBs)
* EDSS Score <3
* Patients covered by health care insurance (social security)
* Written informed consent obtained.
* Onset of symptoms occurring within 60 days of inclusion
* Patients with HIV, HTLV, Hepatitis B, C Syphilis testing negative within 30 days
* Positive EBV serology
* White blood cell count (Leukocytes) > 750/mm3
* Negative pregnancy test

Exclusion Criteria:

* Patients with clinically definite multiple sclerosis
* Patients known to have HIV, HTLV Hepatitis A, B, C or Syphilis infections or patient with active uncontrolled systemic bacterial, viral, parasitic or fungal infections.
* Patients with white blood cell count (Leukocytes) < 750/mm3
* Pregnant or breast feeding women
* Patient with childbearing potentiel refusing efficient contraceptive method
* Patients wishing to be pregnant during the course of the study
* Patients under legal guardianship
* Concomitant participation of any other trial
* Patients with mental or psychiatry condition unable to understand the trial
* Patients with any medically unstable condition or any health conditions that may impact the safety of the patient as determined by the investigator or patient with any stable condition treated with immunotherapy
* Patients with a history of cancer within 5 years or progressive cancer except for basal or cell skin lesions surgically excised and cured, in situ cervical cancer
* Patients unable to comply with protocol.
* Contraindication for MRI or/and any known history of hypersensitivity to contrast medium
* Patients currently treated with immunosuppressive drugs including oral or systemic corticosteroids

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No